CLINICAL TRIAL: NCT03242668
Title: Patient Controlled Paravertebral Analgesia for Video-assisted Thoracoscopic Surgery
Brief Title: Paravertebral Block for Postoperative Analgesia in Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Trung Kien (Other)
Collaborators: Nguyen Truong Giang, PhD. Associate Prof. (Unknown)
Responsible Party: Sponsor-Investigator, Nguyen Trung Kien, Corresponding author,Clinical Research, Vietnam Military Medical University
Organization: Vietnam Military Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103HospitalVMMU
Record Dates: First submitted 2017-07-25; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Pain, Postoperative
Keywords: paravertebral block,PVC,PCA
MeSH Terms: conditions — Pain, Postoperative | interventions — Thoracic Surgery, Video-Assisted; Passive Cutaneous Anaphylaxis; Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: 30 patients, with American Society of Anesthesiologists class I to III risk undergoing elective VATS, aged 32-72 years, scheduled for lung resection surgery , were enrolled in this randomised observer blinded prospective clinical study. Patients who refused to participate, less than 18 years of age, ASA physical status 3 or more, allergy to any of the study drugs, patients having any contraindication for paravertebral block, kyphoscoliosis, presence of acute herpes zoster, chronic pain syndrome, chronic analgesic use and psychiatric disease were excluded from this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PVB using PVC for PCA in VATS (Experimental): The VATS was performed.Paravertebral space was identified by loss of resistance technique combined with video-assisted inside thoracic space before chest close.PVC was inserted.Initiated dose of 0.3ml/kg of Bupivacaine Hydrochloride 1.25mg/ml and Fentanyl Citrate 2 micrograms/ml was administered then continued PCA with background rate 3ml/h, bolus dose 2ml was infused through PVC.
  Interventions: Procedure: VATS; Procedure: PVB using PVC; Drug: PCA

INTERVENTIONS:
Procedure: VATS — General anesthesia was induced with 2.0 mg/kg of propofol, 2.0 mg/kg of fentanyl, and 1.0 mg kg/1 of rocuronium and maintained with continuous infusion 6-12mg/kg/h of propofol,injected 2.0 mg/kg of fentanyl and 0.15 mg/ kg of rocuronium every 30 minutes . All patients were intubated with a double-lumen endobronchial tube for one-lung ventilation.The VATS (Video-Assisted Thoracic Surgery) was performed.
  Other Names: Video-Assisted Thoracic Surgery
Procedure: PVB using PVC — At the end of the surgery, the upper edge of the spinous process of the thoracic vertebral body was recognized. With an epidural needle (Tuohy 22 G; Braun, Melsungen, Germany), the injection point was punctured 2 cm lateral to the midline. The paravertebral space was entered by advancing the Tuohy needle over the superior border of the transverse process. Once in the right place, the PVC was placed through the needle, checking the tip remained placed when removing the needle. The advance of the needle and the entering of the catheter into the paravertebral space were verified all the time by the surgeon using the camera. The PVC (Paravertebral Catheter ) was inserted at this point preversed at this area.
  Other Names: Paravertebral block using paravertebral catheter
Drug: PCA — PVC was inserted.Initiated dose of 0.3ml/kg of Bupivacaine Hydrochloride 1.25mg/ml and Fentanyl Citrate 2 micrograms/ml was administered then continued PCA (Perfusor space pump,Germany)with background rate 3ml/h, bolus dose 2ml was infused through PVC.
  Other Names: Patient controlled analgesia

SUMMARY:
To access the analgesic efficacy of patient controlled thoracic paravertebral analgesia.

DETAILED DESCRIPTION:
The study was carried out on thirty patients who underwent video-assisted thoracic surgery.Paravertebral space was identified by loss of resistance technique under video-assisted inside thoracic space before chest close.Initiated dose of 0.3ml/kg of bupivacaine 0.125%+fentanyl 2 mcg/ml was administered then continued patient-controlled analgesia with background rate 3ml/h, bolus dose 2ml, lockout interval 10 minutes. Postoperative pain was accessed by Visual Analogue Scale at rest and on coughing; monitor the heart rate, blood pressure, respiratory rate, SpO2, arterial blood gas and spirometry in three postoperative consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I to III risk undergoing elective VATS, aged 32-72 years, scheduled for lung resection surgery.

Exclusion Criteria:

* Patients who refused to participate, less than 18 years of age, ASA physical status 3 or more,, allergy to any of the study drugs, patients having any contraindication to placement of PVB, kyphoscoliosis, presence of acute herpes zoster, chronic pain syndrome, chronic analgesic use and psychiatric disease.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
VAS score at rest and on coughing | 72 hours
  Using VAS scale (Atrazennica)

SECONDARY OUTCOMES:
Analgesia effects on respiratory function | three postoperative consecutive days
  Using Spirometry (Chestgraph H1 - 105,Japane) to evaluate respiratory index
Arterial blood gas values | three postoperative consecutive days
  Using Arterial blood gas analysis (STAT Model No.MCP9819-065, Martel Instruments Ltd)
The number dermatome inhibition | three postoperative consecutive days
  Using pin-prick test
Rescue analgesia | three postoperative consecutive days
  When VAS score equal to or more than 4 using fentanyl to manage pain
Patient's satisfaction | three postoperative consecutive days
  Using questionaire with 4 levels :not good,satisfied,good,very good

OTHER OUTCOMES:
Side effects and complications | three postoperative consecutive days
  Respiratory depression (respiratory rate < 8 breaths/min), ,confusion, sedation, urinary retention, nausea, vomiting, headache and pruritus was evaluated.
Heart rate | three postoperative consecutive days
  Using monitoring (Philips)
Blood pressure | three postoperative consecutive days
  Using monitoring (Philips)

CONTACTS AND LOCATIONS:
Locations (1):
- Vietnam Military Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided